CLINICAL TRIAL: NCT02096731
Title: Combined Bronchodilators in Chronic Obstructive Pulmonary Disease and the Risk of Adverse Cardio-pulmonary Events: A Population-based Observational Study
Brief Title: Combined Bronchodilators in Chronic Obstructive Pulmonary Disease and the Risk of Adverse Cardio-pulmonary Events
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.526
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- LABA + tiotropium
- LABA mono
- neither tiotropium nor LABA
- tiotropium + LABA
- tiotropium mono

SUMMARY:
Background: Recent observational studies have reported possible arrhythmogenic effects with long-acting beta-agonists (LABA), while the long-acting anticholinergic tiotropium has been associated with cardiovascular and cerebrovascular events. Finally, pneumonia was the object of a recent signal in trials of LABAs submitted for marketing approval.

Aim: To assess the potential cardio-pulmonary risk arising from the concurrent use of two long-acting bronchodilators as well as from monotherapy use of each of the long-acting bronchodilators.

Methods: A series of population-based cohort studies, using both cohort and nested case-control analyses will be conducted using data from the United Kingdom's Clinical Practice Research Datalink (CPRD). The base cohort will consist of new users of long-acting bronchodilators from Jan 2002 until Aug 2012, age >= 55 with chronic obstructive pulmonary disease (COPD) and at least two years of baseline medical history information. The high-dimensional propensity score technique will be used to match new users of each long-acting bronchodilator and new users of two bronchodilators with comparable subjects from the base cohort, with one-year follow-up for outcomes of acute myocardial infarction, stroke, heart failure, arrhythmia and community acquired pneumonia. Data will be analysed using time-dependent Cox proportional hazard regression models and conditional logistic regression models.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* New users of long-acting bronchodilators, either a LABA or tiotropium, between January 2002 and August 2012
* Age >= 55 years

Exclusion criteria:

- Use of LABA or tiotropium in the two years prior to cohort entry

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of tiotropium or long-acting beta agonists
Sampling Method: Non-Probability Sample
Enrollment: 115397 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The base cohort included 115,397 new users of tiotropium or a LABA (+/- ICS) between 01Jan2002 & 31Aug2013.These patients included 26,442 new users of tiotropium & 88,955 new users of LABA.Patients initiating treatment with both bronchodilators on the same date were excluded.
Pre-assignment Details: Patients receiving combination therapy were those who either added tiotropium to LABA, or added LABA to tiotropium.
  In the Participant Flow & Baseline Characteristics modules, no participants were represented in both the "Tiotropium" & the "LABA" Arms/Groups.
Groups:
- Tiotropium: Participants who were new users of tiotropium.
- LABA: Participants who were new users of a long-acting beta2 agonist (LABA) with or without inhaled corticosteroid (ICS).
Period: Overall Study
Arm/Group | Tiotropium | LABA
Started | 26442 | 88955
Completed | 26442 | 88955
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who were new users of tiotropium or a long-acting beta agonist (LABA) with or without ICS. Estimates based on overall patients before propensity score matching (base cohort).
  New use was defined as a first use of either bronchodilator without use of either drug of interest during the previous two years
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | LABA | Total
Number analyzed (Participants) | 26442 | 88955 | 115397
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (9.0) | 69.4 (9.4) | 69.9 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 11741 | 48912 | 60653
  Male | 14701 | 40043 | 54744

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Infarction
Description: The acute myocardial infarction (MI) rate per 1000 patients per year after matching on high-dimensional propensity score and inhaled corticosteroid (ICS) use in the year prior to cohort entry.
  No. = Number
Time Frame: Up to 12 months
Population: The subset of patients from the base cohort who were either on monotherapy (who stayed on monotherapy) or combination therapy (who added tiotropium to LABA or added LABA to tiotropium) and were matched via propensity score.
Measure: Number; unit: No. of incident MI/1000patients/ year
Groups:
- Monotherapy: Participants remaining on a single long-acting bronchodilator - monotherapy.
- Combination Therapy: Participants who added another long-acting bronchodilator to the previous long-acting bronchodilator (Tiotropium plus LABA+/-ICS) - combination therapy
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 31138 | 31138
No. of incident MI/1000patients/ year | 10.1 | 11.3
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.92 to 1.37] — HR adjusted for 10 year age groups, sex, calendar year of cohort entry, the decile of propensity score, ipratropium use prior to cohort entry and time since entry into base cohort. Ratio calculated as combination therapy divided by monotherapy

2. Primary Outcome: Stroke
Description: The stroke rate per 1000 patients per year after matching on high-dimensional propensity score and inhaled corticosteroid (ICS) use in the year prior to cohort entry.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: No. of incident stroke/1000patients/year
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 31123 | 31123
No. of incident stroke/1000patients/year | 8.3 | 7.0
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.69 to 1.10] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Heart Failure
Description: The heart failure (HF) rate per 1000 patients per year after matching on high-dimensional propensity score and inhaled corticosteroid (ICS) use in the year prior to cohort entry.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: No. of incident HF/1000patients/year
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 31174 | 31174
No. of incident HF/1000patients/year | 29.3 | 33.9
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [1.03 to 1.30] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cardiac Arrhythmia
Description: The cardiac arrhythmia (CA) rate per 1000 patients per year after matching on high-dimensional propensity score and inhaled corticosteroid (ICS) use in the year prior to cohort entry.
Time Frame: Up to 12 months
Population: The subset of patients from the base cohort who were either on monotherapy (who stayed on monotherapy) or combination therapy (who added tiotropium to LABA or added LABA to tiotropium), who can be linked to the Hospital Episode Statistics database, and were matched via propensity score.
Measure: Number; unit: No. of incident CA/1000patients /year
Groups:
- Monotherapy: Participants who can be linked to the Hospital Episode Statistics database and who remained on a single long-acting bronchodilator.
- Combination Therapy: Participants who can be linked to the Hospital Episode Statistics database and who added another long-acting bronchodilator to the previous long-acting bronchodilator.
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 18861 | 18861
No. of incident CA/1000patients /year | 10.0 | 10.7
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.81 to 1.36] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Community Acquired Pneumonia
Description: The community acquired pneumonia rate per 1000 patients per year after matching on high-dimensional propensity score and inhaled corticosteroid (ICS) use in the year prior to cohort entry.
  Pt. = Patient
Time Frame: Up to 12 months
Population: as for outcome 4
Measure: Number; unit: No.of incident Pneumonia/1000 pt./year
Groups:
- Monotherapy: Participants who can be linked to the Hospital Episode Statistics database and who remained on a single long- acting bronchodilator.
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 18867 | 18867
No.of incident Pneumonia/1000 pt./year | 63.0 | 84.6
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.23 to 1.50] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Given the study design, serious and other (non-serious) adverse events were not collected and therefore adverse event data is not presented
Arm/Group | Tiotropium | LABA
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study measures may be subject to misclassification. Diagnoses codes based on read codes and not laboratory or clinical measures. Residual confounding is possible as the analysis is dependent on only recorded information in patients' clinical records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.